CLINICAL TRIAL: NCT04919213
Title: Safer Online Lives: Use of the Internet & Social Media by People With Intellectual Disabilities
Acronym: SOL
Status: Completed | Type: Observational
Sponsor: University of Kent (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 293445
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2021-06

CONDITIONS: Intellectual Disability
Keywords: Intellectual Disability; Internet use; Social Inclusion; Risks; Quality of life; Service provision
MeSH Terms: conditions — Intellectual Disability; Social Inclusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Individuals with Intellectual Disabilities: Individuals will be invited to take part in an online survey (paper version will also be available). The participants will be recruited through advertisements on relevant platforms (e.g., Facebook, Twitter) and through relevant social care organisations. The study hopes to recruit 100 individuals from all over England (UK). A subgroup will be asked if they would like to take part in a one-to-one open-ended interview (n=20) and/or in direct observations (n=30).
- Family carers: Family carers (n=50) of people with intellectual disabilities in England, who use the internet, will be invited to take part in an online survey. A subgroup of family carers (n=7) will be asked if they would like to take part in a focus group.
- Paid carers: Paid carers (n=50) of people with intellectual disabilities in England, who use the internet, will be invited to take part in an online survey. A subgroup of paid carers (n=7) will be asked if they would like to take part in a focus group.
- Professionals with safeguarding responsibilities: Professionals with safeguarding duties (e.g., social workers, learning disability nurses, police and safeguarding adults board members) supporting people with ID in England who use the internet will also be invited to take part in an online survey (n=50). A subgroup (n=7) from London and Kent (England, UK) will be asked if they would like to take part in a focus group.

SUMMARY:
The objective of this study is to explore the benefits of internet use for people with intellectual disabilities (ID), the risks they might come up against while online, the barriers people with ID might come across due to the 'digital divide', and the opportunities offered by being online. The views and experiences of family carers and/or paid carers as well as the views of other safeguarding practitioners will also be investigated.

DETAILED DESCRIPTION:
The most recent estimate is that more than three billion people are using the internet globally and people with ID are not an exception. Children and adults with ID increasingly live in homes with internet access and use the internet to get information about care, health, shopping, accessing social media sites, downloading or watching videos etc.

Benefits of the Internet: Compared to the general population, people with ID are often more likely to have narrow social networks consisting of either other people with disabilities, their families and/or their carers, usually feeling socially isolated and lonely. The internet can help people with ID form and maintain social relationships, but also gain access to expert guidance and information regarding care, health, employment etc.

Online Vulnerabilities: Previous research has identified a link between the use of internet and online risks for both people with and without ID. Such risks include abuse through online dating, being the victim of a fraud etc. Although anyone can be at risk of the above, it has been suggested that such risks are increased when individuals are particularly vulnerable to abuse. Research evidence has demonstrated that people with ID have several negative experiences online such as verbal abuse, sexual exploitation, mistreatment and violence. Furthermore, it has been shown that people with ID who have previous histories of abuse, isolation, and/or depression are more at risk of becoming victims of online sexual exploitation and abuse than others.

Acquiescence and acceptability are also very common in this population. Their desire to "fit in", be liked and willingness to please, might place people with ID in a vulnerable position. Likewise, studies have suggested that the type and severity of an ID, as well as age, could be influencing online risks. For example, people with lower IQ or with lack of social communication skills might have difficulties understanding other people's intentions, which makes them particularly vulnerable to online exploitation, abuse, theft and manipulation.

Existing Evidence: Given that only a very small amount of studies have looked at the internet use and risks for people with ID, there is no study looking at the benefits and opportunities of internet use. Therefore, there is a clear need to investigate this further. Also, all existing studies have focused on small numbers of participants leaving a clear gap in the literature. Only a small number of studies have taken into account family and paid carers' views. Even though the findings derived from these studies cannot be generalised, they act as a useful starting point to highlight the need for further exploration of internet use and online risks for people with ID.

In summary, the purpose of the proposed study is to explore the following four key areas: benefits of using the internet, barriers people with ID face, online risks and online opportunities. The study will also investigate the views (positive and negative) of different stakeholders on the issue; such as family carers, paid carers, safeguarding practitioners, police and people with ID. Furthermore, the proposed study will address the gap in the literature and enhance social care practice by highlighting the importance of providing support for use of internet in order to reduce the current 'digital divide' and also identify areas that future interventions around online safety for people with ID should target.

ELIGIBILITY:
Inclusion Criteria:

* Adults with ID in England who use the internet.
* Carers of people with ID who use the internet.
* Safeguarding professionals working /have worked with people with ID that have been using/have used the internet.
* All participants must be based in England

Exclusion Criteria:

* Participants without an ID / carers of participants without an ID/ safeguarding professionals who have not worked with people with an ID.
* Participants with ID who do not have internet access or chose to not use the internet.
* Participants that do not have the capacity to consent according to the Mental Capacity Act (2005).
* Participants who are not able to communicate verbally will be excluded from the interviews, observations and focus groups; however, they will be included in the questionnaires assessments.
* Carers of people with ID who do not use the internet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with ID who use the internet and carers and professionals who support adults who use the internet.
Sampling Method: Non-Probability Sample
Enrollment: 429 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Online questionnaires - individuals with ID | Through study completion, an average of 18 months
  A questionnaire will be used to investigate the online experiences of adults with ID. Four main key areas will be explored (benefits of using the internet, barriers, risks and opportunities). An easy read adapted version of the Facebook Intensity Scale (FIS; Ellison, Steinfield, & Lampe, 2007) will be used to explore participants' social media usage.
Online questionnaires - family carers, paid carers and safeguarding practitioners | Through study completion, an average of 18 months
  The questionnaire explores the same four key areas as for people with ID (benefits of using the internet for people with ID, barriers, risks and opportunities). A modified version of the questionnaire used in Chadwick et al.'s (2017) study will be used as the basis for the stakeholder's questionnaires.

SECONDARY OUTCOMES:
Observations | Through study completion, an average of 18 months
  The current study will create an app, specifically designed for people with ID. The participants will be given the task to help an avatar and guide their next step on some scenarios. Participants will be presented with multiple scenarios covering the study's four key areas. In total two avatars will be developed (one male and one female) following similar scenarios.
A "think-aloud" observation | Through study completion, an average of 18 months
  The observation will explore the participants' line of thought while online and their reasoning when making decisions. The participant will be asked to talk the researcher through each stage of his/her thinking process and decision making process when online. This observational method is particularly useful for people with ID who may not be very articulate.
Qualitative interviews | Through study completion, an average of 18 months
  20 people with ID who use the internet will be interviewed to collect in depth information and further explore their views on the study's four key areas. The interviews will be conducted once and will be qualitative, semi- structured interviews (with prompts).
Focus groups | Through study completion, an average of 18 months
  The investigators will run 4 separate focus groups. One with family carers, one with paid carers, one with safeguarding practitioners and one including a mixture of paid, family carers and safeguarding practitioners to understand their perspectives and experiences on internet use for people with ID. It is intended that the carers will be independent of the subgroup of people with ID that will take part in the interviews, although there might be some overlaps.

CONTACTS AND LOCATIONS:
Overall Officials: Paraskevi Triantafyllopoulou, PhD, Principal Investigator — University of Kent
Locations (1):
- University of Kent, Canterbury, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blackburn C, Read J. Using the Internet? The experiences of parents of disabled children. Child Care Health Dev. 2005 Sep;31(5):507-15. doi: 10.1111/j.1365-2214.2005.00541.x. PMID 16101645
- [Background] Didden R, Scholte RH, Korzilius H, de Moor JM, Vermeulen A, O'Reilly M, Lang R, Lancioni GE. Cyberbullying among students with intellectual and developmental disability in special education settings. Dev Neurorehabil. 2009 Jun;12(3):146-51. doi: 10.1080/17518420902971356. PMID 19466622
- [Background] Finlay WM, Lyons E. Acquiescence in interviews with people who have mental retardation. Ment Retard. 2002 Feb;40(1):14-29. doi: 10.1352/0047-6765(2002)0402.0.CO;2. PMID 11806730
- [Background] Lough E, Fisher MH. Internet use and online safety in adults with Williams syndrome. J Intellect Disabil Res. 2016 Oct;60(10):1020-30. doi: 10.1111/jir.12281. Epub 2016 May 12. PMID 27174494
- [Background] Molin M, Sorbring E, Lofgren-Martenson L. Teachers' and parents' views on the Internet and social media usage by pupils with intellectual disabilities. J Intellect Disabil. 2015 Mar;19(1):22-33. doi: 10.1177/1744629514563558. Epub 2014 Dec 17. PMID 25524596
- [Background] Normand CL, Sallafranque-St-Louis F. Cybervictimization of Young People With an Intellectual or Developmental Disability: Risks Specific to Sexual Solicitation. J Appl Res Intellect Disabil. 2016 Mar;29(2):99-110. doi: 10.1111/jar.12163. Epub 2015 Apr 13. PMID 25871891
- [Background] Chiner, E., Gómez-Puerta, M., & Cardona-Moltó, M. C. Internet use, risks and online behaviour: The view of internet users with intellectual disabilities and their caregivers. British journal of learning disabilities. 2017; 45(3): 190-197.
- [Background] Chadwick, D. D., Quinn, S., & Fullwood, C. Perceptions of the risks and benefits of Internet access and use by people with intellectual disabilities. British Journal of Learning Disabilities. 2017; 45(1): 21-31.
- [Background] Ellison, B. N., Steinfield, C., & C, L. The Benefits of Facebook "Friends:" Social Capital and College Students' Use of Online Social Network Sites. Journal of Computer-Mediated Communication. 2007; 1143-1168.
- [Background] Forrester-Jones, R., Carpenter, J., Coolen-Schrijner, P., Cambridge, P., Tate, A., Beecham, J., ... & Wooff, D. The social networks of people with intellectual disability living in the community 12 years after resettlement from long-stay hospitals. Journal of Applied Research in Intellectual Disabilities. 2006; 19(4): 285-295.
- [Background] Gravell, C. 2012. Loneliness and cruelty: people with learning disabilities and their experience of harassment, abuse and related crime in the community. London: Lemos and Crane.
- [Background] Gutiérrez P, Martorell A. People with intellectual disability and ICTs. Rev. Comun. 2011; 36: 173-180.
- [Background] Holmes KM, O'Loughlin N. The experiences of people with learning disabilities on social networking sites. British Journal of Learning Disabilities. 2012; 42(1): 1-5.
- [Background] Kirwan G, Power A. 2013. Cybercrime: The psychology of online offenders. Cambridge: University Press.
- [Background] Löfgren-Mårtenson L. Love in cyberspace: Swedish young people with intellectual disabilities and the Internet. Scandinavian Journal of Disability Research. 2008; 10(2): 125-138.
- [Background] Lussier-Desrochers D, Normand CL, Romero-Torres A, Lachapelle Y, Godin-Tremblay V, Dupont MÈ, ... & Bilodeau P. Bridging the digital divide for people with intellectual disability. Cyberpsychology: Journal of Psychosocial Research on Cyberspace. 2017; 11(1).
- [Background] Meeker M, Wu L. 2018. Internet trends 2018 (Code 2018). Retrieved from https://www.businessinsider.com/mary-meeker-internet-trends-2018-full-slide-deck-2018-5?r=US&IR=T
- [Background] Sallafranque-St-Louis F, Normand CL. From solitude to solicitation: How people with intellectual disability or autism spectrum disorder use the internet. Cyberpsychology: Journal of Psychosocial Research on Cyberspace. 2017; 11(1).
- [Background] Steinfield C, Ellison NB, Lampe C. Social capital, self-esteem, and use of online social network sites: A longitudinal analysis. Journal of Applied Developmental Psychology. 2008; 29(6): 434-445.
- See also: Research Project homepage — https://research.kent.ac.uk/tizard/safer-online-lives/